CLINICAL TRIAL: NCT01109433
Title: Immunogenetic Mechanisms in Behcet's Disease
Status: Terminated | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100093; 10-EI-0093
Record Dates: First submitted 2010-04-22; First posted 2010-04-23 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2018-12-17

CONDITIONS: Behcet's Disease; Uveitis
Keywords: Behcet's Disease; Intermediate Uveitis; Uveitis; Immunogenetics
MeSH Terms: conditions — Behcet Syndrome; Uveitis; Uveitis, Intermediate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Background:

- Uveitis, the inflammation of the interior of the eye, is responsible for numerous new cases of legal blindness every year. Uveitis can be caused by Beh(SqrRoot)(Beta)et s disease (BD), a chronic inflammatory disorder that can affect the eye, mucous membranes, and other body organs such as the joints, intestinal tract, blood vessels, and central nervous system.

Objectives:

The purpose of this study is to see how genes affect Beh(SqrRoot)(Beta)et s disease and if there are differences in Beh(SqrRoot)(Beta)et s disease among people of different backgrounds.

Eligibility:

* Individuals who have a diagnosis of BD and are enrolled in another NIH study.
* Individuals who are willing to donate blood for the purposes of this research study and who are willing to have their blood stored for possible future/other research purposes.

Design:

* As part of the study, blood samples will be drawn from participants when an exacerbation in disease activity occurs and before and after any significant change in treatment for BD.
* No treatments will be provided in this study.

DETAILED DESCRIPTION:
Uveitis is responsible for approximately 30,000 cases of new legal blindness in the United States and 2.8-10% of all cases of blindness. Beh(SqrRoot)(Beta)et s disease (BD) is a chronic relapsing multisystem inflammatory disorder of unknown etiology that is characterized by intraocular inflammation, oral and mucosal ulcerations, cutaneous lesions and inflammation that may affect other body organs such as the joints, intestinal tract, epididymis, blood vessels and the central nervous system (2). The need for a safer and more effective therapy for patients with ocular manifestations of BD refractory to or intolerant of systemic immunosuppressive therapy warrants further investigation. Reports define a specific role for interleukin (IL)-17A in the pathogenesis of Beh(SqrRoot)(Beta)et s disease.

This protocol will evaluate immune mediators including cytokine profiles (soluble and intracellular), lymphocyte phenotyping and regulatory T-cells in participants with BD. Epigenetic modifications will also be studied.

Additionally, it has been suggested that American/Western BD patients may have different disease characteristics than their Mediterranean counterparts. The disease characteristics of American/Western and Mediterranean BD patients will be compared and evaluated. Blood samples from BD participants that have participated in other NIH protocols where participants consented for other or future use of samples has been obtained will be collected (particularly from current participants of NIH protocol 03-AR-0173 in which NEI is a collaborator). In summary, the results will be analyzed with respect to disease in different ethnic groups, and clinical features of the disease (e.g., ocular vs. non-ocular involvement, active vs. quiescent disease).

Anonymous blood samples (matched for race, age and sex) will be obtained from the NIH clinical center (CC) blood bank and will be compared to the diseased samples.

ELIGIBILITY:
* INCLUSION CRITERIA:

One of the following must be true:

* Participants must have a diagnosis of BD according to the International Study Group for BD criteria or modified Japanese criteria, be enrolled in another NIH study and be willing to donate their blood for the purposes of this research study.
* Participants must be willing to have their blood stored for future/other research.

EXCLUSION CRITERIA:

Eligible participants who do not wish to donate their blood sample or undergo a blood draw for the purposes of this research study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-04-15; Study Completion 2018-12-17

PRIMARY OUTCOMES:
Establishing evidence for serum biomarkers associated with BD and establishing demethylation differences between ocular and non-ocular BD participants and controls. | Ongoing

SECONDARY OUTCOMES:
To explore associations between disease severity and treatment response with observed epigenetic modifications and biomarkers. | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Hatice N Sen, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gritz DC, Wong IG. Incidence and prevalence of uveitis in Northern California; the Northern California Epidemiology of Uveitis Study. Ophthalmology. 2004 Mar;111(3):491-500; discussion 500. doi: 10.1016/j.ophtha.2003.06.014. PMID 15019324
- [Background] Chamberlain MA. Behcet's syndrome in 32 patients in Yorkshire. Ann Rheum Dis. 1977 Dec;36(6):491-99. doi: 10.1136/ard.36.6.491. PMID 596943
- [Background] Jankowski J, Crombie I, Jankowski R. Behcet's syndrome in Scotland. Postgrad Med J. 1992 Jul;68(801):566-70. doi: 10.1136/pgmj.68.801.566. PMID 1437955